CLINICAL TRIAL: NCT05891678
Title: The Value of Doppler Study of Central Retinal Artery in Diagnosis of Increased ICP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Inas Ahmed Sayed Ammar (Other)
Responsible Party: Sponsor-Investigator, Inas Ahmed Sayed Ammar, Head of intensive care unit, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRA doppler in increased ICP
Record Dates: First submitted 2023-03-03; First posted 2023-06-07 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Increased Intracranial Pressure
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (N) (No Intervention): Central retinal artery Doppler in patient with normal ICP
- Intervention group (H) (Active Comparator): Central retinal artery Doppler in patient with increased ICP
  Interventions: Radiation: doppler study of central retinal artery

INTERVENTIONS:
Radiation: doppler study of central retinal artery — pulsed wave Doppler after decreasing the sample volume to fit inside the center of CRA. We will measure the peak systolic velocity (PSV), end diastolic velocity (EDV), and the resistivity index which equal PSV-EDV/PSV, we will measure 3 times and the expected normal value is less than 0.7.
  Arms: Intervention group (H)

SUMMARY:
The purpose of this study is to evaluate the diagnostic value of central retinal artery Doppler study in case of increased intracranial pressure.

DETAILED DESCRIPTION:
In neurocritical care, the detection of raised intracranial pressure (ICP) remains crucial as it is associated with poor outcome . Invasive ventricular devices are the gold standard for continuous and reliable measurement of ICP however their placement could be challenging due to blood coagulation disorder or lack of surgical availability. Moreover, malfunction or obstruction of ventricular catheters has been reported to occur as often as 6%. Recently Julie.et al. revealed in his met analysis that optic nerve sheath diameter (ONSD) has a good level of diagnostic accuracy for detecting intracranial hypertension with a pooled sensitivity of 0.9. The central retinal artery (CRA) is an end artery branch of the internal carotid artery that joins the optic nerve 1cm behind the globe and enters the retina on the optic nerve head . Central retinal artery is located inside the optic nerve sheath, and The optic nerve is part of the central nervous system and the intraorbital subarachnoid space surrounding the optic nerve is subject to the same pressure changes as the intracranial compartment,so we should expect any increase of ICP will compress the central retinal artery exactly the same as basal cerebral arteries. Central retinal artery circulation is low resistance circulation with good diastolic flow and upper limit of resistivity index is 0.7. So, any compression of CRA will decrease the diastolic flow and increase RI. Kamil.et al. studied the blood flow velocity changes in orbital arteries by using Doppler sonography in eight patients with brain death and increased ICP. Peak systolic and end-diastolic velocities and resistive indices of the ophthalmic and central retinal arteries were evaluated. they observed the absence or reversal of end diastolic blood flow in these arteries. If the intracranial pressure is higher than the end-diastolic pressure of the cerebral arteries diastolic flow reversal occurs. If the intracranial pressure exceeds systolic pressure blood flow is entirely ceased with complete and irreversible loss of brain function CRA is a superficial, easy accessible without bony obstacle like transcranial doppler (TCD) and the learning curve of its Doppler study can be very steep, so it could has a big role in management of cases with increased ICP.

ELIGIBILITY:
Inclusion Criteria:

* All Patients with cerebral stroke either ischemic or hemorrhagic
* All Patients with traumatic brain injury including those on mechanical ventilation

Exclusion Criteria:

* Patients with eye trauma
* Patients with either arteritic or non arteritic central retinal artery occlusion

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Central retinal artery resistivity index | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Central retinal artery resistivity index computed by PSV (cm/s ) and EDV (cm/s) reflects vascular resistance peripheral to the measuring location. The present study evaluate the correlation of Central retinal artery resistive index with increased intracranial pressure .
peak systolic velocity ( cm/s) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  on a doppler waveform PSV correspond to each tall "peak " in the spectrum window calculated by build in software
end diastolic velocity ( cm/s ) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  on a doppler waveform EDV correspond to the point marked at the end of the cardiac cycle calculated by build in software

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Kas AL- Ainy Fuculty of medicine, Cairo, Egypt